CLINICAL TRIAL: NCT04744610
Title: Prospective Self-controlled Study for Shortening the Time Before Taking Delayed Radiographs With Iodized Oil Hysterosalpingography
Brief Title: Self-controlled Study Between 4-hour and 24-hour Delayed Radiographs in HSG Using OSCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-20200261-R
Record Dates: First submitted 2021-01-06; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Infertility
Keywords: Infertility; Hysterosalpingography; Oil-soluble contrast medium
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-hour delayed radiographs (Other): The follow-up radiographs was taken 4 h after the HSG operation.
  Interventions: Diagnostic Test: Add 4-hour delayed radiographs

INTERVENTIONS:
Diagnostic Test: Add 4-hour delayed radiographs — Normal patients only need to take delayed radiographs 24h after HSG operation. In this study, 4-hour delayed radiographs were added to the 24-hour delayed radiographs, so that the patients had to take one more delayed radiographs .

SUMMARY:
Background of the study:

Hysterosalpingography (HSG) is widely used for the female infertility workup. Many studies have demonstrated that the use of oil-soluble contrast medium (OSCM) ethiodized oil for HSG surgery can improve pregnancy rates. However,The 24-hour delayed radiographs of OSCM HSG also brought some inconvenience to the patients , for example, patients need to make two trips to the hospital.

Objective of the study:

The purpose of this study was to compare OSCM HSGs using 4-hour and 24-hour delayed radiographs in terms of diagnosing tubal patency and identifying the presence of pelvic adhesions.

Study design:

Prospective, open label, self - controlled study

Study population:

Infertile patients scheduled for an OSCM HSG

ELIGIBILITY:
Inclusion Criteria:

* Having spontaneous ovulation or inducing ovulation;
* Infertility lasting for 12 months;
* Conforms to the indications of hysterosalpingography;
* Understand and sign the informed consent;

Exclusion Criteria:

* Iodine allergy or hyperthyroidism
* Acute genital tract inflammation or abnormal leucorrhea examination;
* Abnormal vaginal bleeding;
* Fever or preoperative temperature higher than 37.5℃ within 3 days before angiography;
* Severe insufficiency of cardiopulmonary or liver function;
* During pregnancy and menstruation;
* With complications that may cause subjects to be unable to follow the study plan or even endanger the patient's safety or social environment;
* Patients who are participating in other clinical studies or who are not suitable for inclusion in this study due to other reasons considered by the researchers.

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Difference in diagnosis of fallopian tube patency between 4 hours delayed radiographs and 24 hours delayed radiographs. | The evaluation was performed within 1 day after completion of the 24 hours delayed radiographs.
  The diagnostic results of 4 hours delayed radiographs and 24 hours delayed radiographs were evaluated by two radiologists with more than 5 years' working experience. In case of any dispute, the two doctors reached an agreement after discussion.
  The results were defined as : completely consistent; mostly consistent;partly consistent;completely different.

SECONDARY OUTCOMES:
Difference in the diagnosis of patency of proximal fallopian tube between 4 hours delayed radiographs and 24 hours delayed radiographs | The evaluation was performed within 1 day after completion of the 24 hours delayed radiographs.
  The diagnostic results of 4 hours delayed radiographs and 24 hours delayed radiographs were evaluated by two radiologists with more than 5 years' working experience. In case of any dispute, the two doctors reached an agreement after discussion.
  The results were defined as : completely consistent; mostly consistent;partly consistent;completely different.
Difference in the diagnosis of patency of distal fallopian tube between 4 hours delayed radiographs and 24 hours delayed radiographs | The evaluation was performed within 1 day after completion of the 24 hours delayed radiographs.
  The diagnostic results of 4 hours delayed radiographs and 24 hours delayed radiographs were evaluated by two radiologists with more than 5 years' working experience. In case of any dispute, the two doctors reached an agreement after discussion.
  The results were defined as : completely consistent; mostly consistent;partly consistent;completely different.
Difference in the diagnosis of pelvic lesions between 4 hours delayed radiographs and 24 hours delayed radiographs. | The evaluation was performed within 1 day after completion of the 24 hours delayed radiographs.
  The diagnostic results of 4 hours delayed radiographs and 24 hours delayed radiographs were evaluated by two radiologists with more than 5 years' working experience. In case of any dispute, the two doctors reached an agreement after discussion.
  The results were defined as : completely consistent; mostly consistent;partly consistent;completely different.

OTHER OUTCOMES:
The incidence of adverse events and serious adverse events. | Within one month after hysterosalpingography procedure.
  Adverse event levels were assessed according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Zhu, Study Chair — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No